CLINICAL TRIAL: NCT02233361
Title: Use of Hearing Aids. Development and Implementation of a Counselling Program for Hearing Aid Users.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013/2/0252
Record Dates: First submitted 2014-08-13; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Presbyacusis
Keywords: Hearing rehabilitation; Elderly; Hearing aid use
MeSH Terms: conditions — Presbycusis | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Experimental): The intervention group will be informed in advance of a follow-up appointment six month after they have received their hearing aid. They will know that support will be given and time-use of the hearing aid will be checked out. Counseling on hearing aid use will be given.
  Interventions: Behavioral: Counseling
- Counselling (No Intervention): The control group will not receive any information of a follow-up appointment. However, they will receive a notice on this after six month.

INTERVENTIONS:
Behavioral: Counseling — A randomized controlled design will determine whether hearing aid users who are informed in advance of a follow-up appointment have a different pattern of hearing aid use than a control group that is not preinformed in advance.
  Arms: Counseling

SUMMARY:
The proportion of elderly people is expected to increase greatly within the next couple of decades, resulting in a proportional increase in the need for hearing rehabilitation. However, studies suggest that as many as 40% of hearing aids are never or seldom used. Thus, a major challenge for audiological rehabilitation is facilitating the use of fitted hearing aids.

This study has four objectives; 1) to evaluate the effect of advanced notice of a follow-up appointment on hearing aid use, 2) to implement a specialized counselling program based on MI, 3) to identify barriers to hearing aid use, and 4) to objectively assess hearing aid use with datalogging technology.

DETAILED DESCRIPTION:
Hearing impairment is one of the most common health issues among adults in Western countries. Socioeconomic status and level of family support are known to influence help-seeking among older hearing-impaired individuals. Although hearing loss can have significant adverse effects on an individual's quality of life, these effects have been found to be reversible through the use of hearing aids. Even short-time use has been found to improve the emotional and social experience of hearing impaired subjects. Unfortunately, of the approximately 200 000 people who have been provided with hearing aids in Norway, it is estimated that as many as 20-40% seldom or never use them. Lack of follow-up support and low motivation may explain why hearing impaired people do not use their hearing aids, but few research studies have addressed these issues.

The aim of this study is to evaluate two approaches for increasing hearing aid use, to obtain objective estimates of actual hearing aid use, to identify factors barriers to regular use and to study hearing aid use related to age and gender. The study will examine the extent to which follow-up appointments motivate use of hearing aids among people with hearing loss. A randomized controlled design will determine whether hearing aid users who are informed in advance of a follow-up appointment have a different pattern of hearing aid use than a control group that is not preinformed of the follow-up appointment. For decades, the use of hearing aids has been estimated using questionnaires. In the present study, hearing aid use will be objectively measured in hours pr.day using the hearing aid's datalogging. In addition, the study will develop, implement and evaluate a specialized counseling program for hearing aid users. Difficulties with and barriers to hearing aid use will be documented and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 + years old
* Subjective and objective need for hearing aids.

Exclusion Criteria:

* Not being able to communicate in Norwegian.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The effect of follow-up appointments on hearing aid use | 1 year
  The counseling utilize Motivational Interviewing (MI) to promote hearing aid use. Datalogging will be used to assess changes in hearing aid use.

SECONDARY OUTCOMES:
Hearing aid use measured with datalogging technology | When signed for the hearing aid and six month later
  The use of datalogging technology will strengthen the evaluation by providing an objective measure of hearing aid use. Real time use of hearing aids in hours per day will be assessed by connecting the instrument to the programming tool, Noah.

OTHER OUTCOMES:
Factor Barriers to hearing aid use | At the follow up appointment. Six month after the hearing aid was assigned for.
  Difficulties with and barriers to hearing aid use will be documented and analyzed. Problems and barriers associated with hearing aid use will be recorded and categorized by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Solheim, Ph.d., Principal Investigator — Lovisenberg Diakonale Hospital
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway